CLINICAL TRIAL: NCT07359053
Title: MAGNATE-S: A Phase 2 Exploratory Study of Paclitaxel Polymer Micelles Combined With Gemcitabine and Anti-Angiogenic TKIs (Lenvatinib or Anlotinib) for Advanced Bone and Soft Tissue Sarcomas
Brief Title: MAGNATE-S: Paclitaxel Polymer Micelles Combo in Advanced Sarcoma
Acronym: MAGNATE-S
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Shen Zan, The Director of of the Department of Medical Oncology, Shanghai 6th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-206; 2025-206 (Other: shanghai sixth people's hospital affiliated to shanghai jiao tong university school of medicine)
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Sarcoma
Keywords: advanced sarcoma; Paclitaxel Polymer Micelles
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; lenvatinib; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bone sarcoma (Experimental)
  Interventions: Drug: Paclitaxel Polymer Micelles + Gemcitabine + Lenvatinib
- soft tissue sarcoma (Experimental)
  Interventions: Drug: Paclitaxel Polymer Micelles + Gemcitabine + Anlotinib

INTERVENTIONS:
Drug: Paclitaxel Polymer Micelles + Gemcitabine + Lenvatinib — 1. Paclitaxel Polymer Micelles + Gemcitabine: Paclitaxel Micelles: 230 mg/m² (C1), then 300 mg/m² if tolerated, IV (≥3h), D8, Q3W. Gemcitabine: 800 mg/m², IV (90min), D1&D8, Q3W. Planned for 6 cycles, may extend >6 cycles (based on investigator assessment of continued clinical benefit and patient tolerance) with patient self-pay for Paclitaxel Micelles.
  2. Lenvatinib (Bone Sarcoma): 12-16 mg daily (8-12 mg if <60 kg), continuous oral dosing until progression.
  General Rules: Dose adjustments based on CTCAE v5.0. For patients with systemic benefit (PR/SD per RECIST 1.1 for ≥2 cycles), localized interventions (e.g., surgery, radiation) are permitted following MDT evaluation and with protocol-defined study drug adjustments.
  Arms: bone sarcoma
Drug: Paclitaxel Polymer Micelles + Gemcitabine + Anlotinib — 1. Paclitaxel Polymer Micelles + Gemcitabine: Paclitaxel Micelles: 230 mg/m² (C1), then 300 mg/m² if tolerated, IV (≥3h), D8, Q3W. Gemcitabine: 800 mg/m², IV (90min), D1&D8, Q3W. Planned for 6 cycles, may extend >6 cycles (based on investigator assessment of continued clinical benefit and patient tolerance) with patient self-pay for Paclitaxel Micelles.
  2. Anlotinib (Soft Tissue Sarcoma): 12 mg daily (8 mg if <45 kg), oral (2 wks on/1 wk off) until progression.
  General Rules: Dose adjustments based on CTCAE v5.0. For patients with systemic benefit (PR/SD per RECIST 1.1 for ≥2 cycles), localized interventions (e.g., surgery, radiation) are permitted following MDT evaluation and with protocol-defined study drug adjustments.
  Arms: soft tissue sarcoma

SUMMARY:
What is this study about? This is a medical research study testing a new drug combination ("Paclitaxel Polymer Micelles" + "Gemcitabine" + "Targeted Therapy") for patients with locally advanced unresectable or metastatic bone and soft tissue sarcomas whose disease has progressed after first-line standard therapy. Currently, there is a lack of highly effective subsequent treatment options for these patients.

Why is this study being done? To improve efficacy: the investigators hope this drug combination can control tumor growth more effectively than current treatments.

To reduce toxicity: The "Paclitaxel Polymer Micelles" used in the study is a new formulation that may be safer than traditional paclitaxel, with a lower risk of severe allergic reactions.

For precise treatment: the investigators will select different targeted drugs (Lenvatinib for bone sarcoma or Anlotinib for soft tissue sarcoma) based on the tumor type, aiming for more tailored therapy.

How will the study be conducted?

Design: This is an exploratory study, planning to enroll approximately 46 patients in total, divided into two separate groups (23 for bone sarcoma, 23 for soft tissue sarcoma).

Process: Eligible and consenting patients will receive periodic combined drug therapy. Doctors will regularly evaluate efficacy and monitor safety through blood tests, US, CT, or MRI scans.

Primary Goal: The main focus is to see how many patients experience significant tumor shrinkage (Objective Response Rate), and to record all adverse reactions that occur.

Biomarker Research: To better understand treatment mechanisms and identify potential predictive markers, this study includes the collection of biological samples for future research, with careful design to minimize additional burden. Small extra blood samples will be collected during scheduled routine blood draws required for clinical monitoring. If a tumor biopsy or surgery is performed as part of necessary clinical care, the investigators will request permission to preserve a portion of the remaining tissue that would otherwise be discarded. These samples may be analyzed using techniques such as genetic or protein testing.

What does this mean for participants?

Potential Benefits: Participants have the opportunity to receive the new drug "Paclitaxel Polymer Micelles" free of charge and may benefit from it. Their participation will provide valuable treatment experience for all future patients with similar conditions.

Potential Risks: The drug combination may increase the risk of certain side effects, such as fatigue, nausea, high blood pressure, hand-foot skin reactions, or decreased blood cell counts. The research team has developed detailed plans to prevent and manage these situations.

Voluntary Principle: Participation is completely voluntary. Patients have the right to withdraw from the study at any time, for any reason, without affecting their right to receive other routine medical care.

In summary, this study explores a regimen combining a novel nano-drug, chemotherapy, and precise targeted therapy, aiming to find a more effective and safer treatment option for patients with advanced bone and soft tissue sarcomas who have failed first-line treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent: The subject has signed the informed consent form after receiving and understanding full explanation regarding the trial's purpose, procedures, anticipated efficacy, pharmacological actions, and risks.
* Target Population:

  1. Histologically confirmed advanced/metastatic bone or soft tissue sarcoma. (If recurrence or metastasis is not definitive, a biopsy with frozen section is recommended. Enrollment may proceed if frozen pathology suggests recurrence/metastasis.)
  2. At least one measurable lesion per RECIST 1.1 criteria.
  3. Disease progression after prior first-line standard chemotherapy; ECOG performance status 0-2.
  4. Life expectancy ≥ 3 months.
  5. Willing and able to comply with study procedures, treatment, and follow-up.
  6. No contraindications to paclitaxel polymer micelles, gemcitabine, or small-molecule anti-angiogenic targeted agents.
* Physical Examination and Laboratory Results:

  1. Adequate hematologic function: i) Absolute neutrophil count (ANC) ≥ 1.8 × 10⁹/L; ii) Platelet count ≥ 100 × 10⁹/L; iii) Hemoglobin ≥ 90 g/L. (If transfusions are given during screening, a repeat test after 1 week must meet these criteria.)
  2. Adequate hepatic function: i) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); ii) AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases are present); Alkaline phosphatase (ALP) ≤ 5 × ULN (liver mets) or ≤ 10 × ULN (bone mets).
  3. Adequate renal function: Serum creatinine ≤ 1.5 × ULN or calculated creatinine clearance ≥ 50 mL/min.
  4. Adequate coagulation: INR ≤ 1.5 × ULN and PT/aPTT ≤ 1.5 × ULN, unless on stable anticoagulant therapy.
* Hepatitis B: Subjects positive for HBsAg are eligible if, in the investigator's judgment, their chronic hepatitis B is stable and does not increase the subject's risk.
* Cardiac Function: No symptomatic cardiac insufficiency at baseline (NYHA class ≤ II) and no clinically significant ECG abnormalities.
* Age and Reproductive Status:

  1. Aged 12-70 years (male and female).
  2. Subjects of childbearing potential must agree to use effective contraception during the trial. A negative serum or urine pregnancy test within 24 hours before chemotherapy is required for women of childbearing potential.
  3. Female subjects must not be breastfeeding.

Exclusion Criteria:

* Known allergy or intolerance to any component or excipient of the investigational products.
* Primary brain tumor or central nervous system (CNS) metastases (including leptomeningeal metastases), except for a single, well-controlled, asymptomatic brain metastasis. CNS tumors still presenting with increased intracranial pressure or neuropsychiatric symptoms after treatment.
* Uncontrolled acute or chronic infections, or other severe concurrent medical conditions.
* History of other malignancies within the past 5 years, except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix.
* Active hepatitis or hepatic tumor burden exceeding 50% of the total liver volume.
* Uncontrolled third-space fluid accumulation not manageable by drainage (e.g., moderate to large pleural effusion, pericardial effusion, or ascites). Minimal asymptomatic fluid not requiring intervention may be allowed upon strict review.
* Psychiatric illness or cognitive impairment leading to poor compliance or inability to cooperate and report treatment responses.
* Severe organic disease or major organ failure (e.g., decompensated heart or lung failure) precluding tolerance to chemotherapy.
* Coagulopathy (INR >1.5, APTT >1.5 × ULN), bleeding tendency (e.g., active gastric ulcer, stool occult blood [++], hematemesis and/or melena within the past 3 months, hemoptysis), or tumor proximity to major blood vessels.
* Coronary artery disease above grade I, arrhythmia (including QTc interval >450 ms for males, >470 ms for females), use of antiarrhythmic medication, or relevant underlying cardiac disease/cardiac insufficiency.
* Renal insufficiency, history of renal disease, or proteinuria (urine protein ≥2+ or 24-hour urine protein >1.0 g).
* History of organ transplantation.
* History of substance abuse, chronic alcoholism, or infectious diseases such as AIDS.
* Long-term use of corticosteroids or immunosuppressants.
* Vaccination with live or attenuated vaccines (e.g., measles, mumps, rubella, varicella, yellow fever, rabies, BCG, oral typhoid) within 4 weeks prior to enrollment, or planned vaccination during the study. COVID-19 vaccination is permitted.
* Active hepatitis B (HBV DNA ≥1×10⁴ copies/mL or ≥2000 IU/mL) or hepatitis C (HCV RNA ≥15 IU/mL) infection; positive HIV antibody (unless clinically indicated); or positive syphilis antibody (TPPA).
* Any other condition deemed by the investigator to prevent completion of the trial or render the subject unsuitable (e.g., tumors like GIST or ALK-mutant inflammatory myofibroblastic tumor unsuitable for this chemotherapy regimen).

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | assessed up to 1 year

SECONDARY OUTCOMES:
Progression-Free-Survival | assessed up to 1 year
Disease Control Rate | assessed up to 1 year
Duration of Response | assessed up to 1 year
Time To Progression | assessed up to 1 year
Incidence of adverse events | assessed up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth Peolple'S Hospital, Shanghai, CH, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication of this trial (including de-identified demographic, clinical, efficacy, and safety data), the study protocol, statistical analysis plan, and informed consent form will be made available.
  Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal that has been approved by an independent review committee. Proposals should be directed to the corresponding author.
  Time Frame: Data will become available 12 months after the primary results publication and will remain accessible for 5 years.
  Mechanism: Data will be provided in a secure, de-identified format via a trusted data repository or upon direct request, subject to a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data that underlie the results reported in the primary publication of this trial (including de-identified demographic, clinical, efficacy, and safety data), the study protocol, statistical analysis plan, and informed consent form will be made available.
  Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal that has been approved by an independent review committee. Proposals should be directed to the corresponding author.
  Time Frame: Data will become available 12 months after the primary results publication and will remain accessible for 5 years.
  Mechanism: Data will be provided in a secure, de-identified format via a trusted data repository or upon direct request, subject to a data sharing agreement.
Access Criteria: Individual participant data that underlie the results reported in the primary publication of this trial (including de-identified demographic, clinical, efficacy, and safety data), the study protocol, statistical analysis plan, and informed consent form will be made available.
  Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal that has been approved by an independent review committee. Proposals should be directed to the corresponding author.
  Time Frame: Data will become available 12 months after the primary results publication and will remain accessible for 5 years.
  Mechanism: Data will be provided in a secure, de-identified format via a trusted data repository or upon direct request, subject to a data sharing agreement.